CLINICAL TRIAL: NCT03811574
Title: Effect and Safety of Semaglutide Once-weekly in East Asian Subjects With Overweight or Obesity
Brief Title: STEP 6: Research Study Investigating How Well Semaglutide Works in People Living With Overweight or Obesity
Acronym: STEP 6
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9536-4382; U1111-1201-1629 (Other: World Health Organization (WHO))
Record Dates: First submitted 2019-01-18; First posted 2019-01-22 (Actual); Results first posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-02

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Semaglutide 2.4 mg (Experimental): Participants will receive semaglutide injections once-weekly for 68 weeks. Participants will be initiated at a once-weekly dose of 0.25 mg and follow a fixed-dose escalation regimen, with dose increases every 4 weeks (to doses of 0.5, 1.0, 1.7 and 2.4 mg/week), until the target dose (2.4 mg) is reached after 16 weeks. Participants will continue semaglutide 2.4 mg until week 68.
  Interventions: Drug: Semaglutide
- Placebo (semaglutide 2.4 mg) (Placebo Comparator): Participants will receive placebo (semaglutide) injections once-weekly for 68 weeks. Participants will be initiated at a once-weekly dose of 0.25 mg and follow a fixed-dose escalation regimen, with dose increases every 4 weeks (to doses of 0.5, 1.0, 1.7 and 2.4 mg/week), until the target dose (2.4 mg) is reached after 16 weeks. Participants will continue placebo (semaglutide 2.4 mg) until week 68.
  Interventions: Drug: Placebo (semaglutide)
- Semaglutide 1.7 mg (Experimental): Participants will receive semaglutide injections once-weekly for 68 weeks. Participants will be initiated at a once-weekly dose of 0.25 mg and follow a fixed-dose escalation regimen, with dose increases every 4 weeks (to doses of 0.5, 1.0 and 1.7 mg/week), until the target dose (1.7 mg) is reached after 12 weeks. Participants will continue semaglutide 1.7 mg until week 68.
  Interventions: Drug: Semaglutide
- Placebo (semaglutide 1.7 mg) (Placebo Comparator): Participants will receive placebo (semaglutide) injections once-weekly for 68 weeks. Participants will be initiated at a once-weekly dose of 0.25 mg and follow a fixed-dose escalation regimen, with dose increases every 4 weeks (to doses of 0.5, 1.0 and 1.7 mg/week), until the target dose (1.7 mg) is reached after 12 weeks. Participants will continue placebo (semaglutide 1.7) until week 68.
  Interventions: Drug: Placebo (semaglutide)

INTERVENTIONS:
Drug: Semaglutide — Semaglutide injections will be administered once-weekly by a pre-filled pen-injector at the same day of the week (to the extent possible). Injections may be administered in the thigh, abdomen or upper arm, at any time of day irrespective of meals.
  Arms: Semaglutide 1.7 mg; Semaglutide 2.4 mg
Drug: Placebo (semaglutide) — Placebo (semaglutide) injections will be administered once-weekly by a pre-filled pen-injector at the same day of the week (to the extent possible). Injections may be administered in the thigh, abdomen or upper arm, at any time of day irrespective of meals.
  Arms: Placebo (semaglutide 1.7 mg); Placebo (semaglutide 2.4 mg)

SUMMARY:
This study will look at the change in participants' body weight from the start to the end of the study. This is to compare the effect on body weight in people taking semaglutide (a new medicine) and people taking "dummy" medicine. In addition to taking the medicine, participants will have talks with study staff about healthy food choices, how to be more physically active and what participants can do to lose weight. Participants will either get semaglutide or "dummy" medicine - which treatment participants get is decided by chance. Participants are three times as likely to get semaglutide as "dummy" medicine. Participants will need to take 1 injection once a week. The study medicine is injected with a thin needle in a skinfold in the stomach, thigh or upper arm. The study will last for about one and a half years. Participants will have 14 clinic visits and 11 phone calls with the study doctor.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age more than or equal to 18 years at the time of signing informed consent
* BMI more than or equal to 27.0 kg/m^2 with more than or equal to 2 weight related comorbidities (treated or untreated) or BMI more than or equal to 35.0 kg/m^2 with more than or equal to 1 weight related comorbidity (treated or untreated) according to the JASSO guideline. At least one comorbidity should be hypertension or dyslipidaemia (Japan only: or T2D)
* History of at least one self-reported unsuccessful dietary effort to lose body weight
* For subjects with T2D at screening (Japan only): a) Diagnosed with T2D more than or equal to 180 days prior to the day of screening. b) HbA1c 7.0-10.0% (53-86 mmol/mol) (both inclusive)

Exclusion Criteria:

* A self-reported change in body weight more than 5 kg (11 lbs) within 90 days before screening irrespective of medical records
* For subjects without T2D at screening: HbA1c more than or equal to 48 mmol/mol (6.5%) as measured by the central laboratory at screening
* For subjects with T2D at screening (Japan only): a) Renal impairment measured as estimated glomerular filtration rate (eGFR) value of less than 30 mL/min/1.73 m^2 (less than 60 mL/min/1.73 m^2 in subjects treated with sodium-glucose co-transporter 2 inhibitor (SGLT2i)) according to chronic kidney disease epidemiology (CKD-EPI) creatinine equation as defined by kidney disease improving global outcome (KDIGO) 2012 by the central laboratory at screening. b) Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a pharmacologically pupil-dilated fundus examination performed by an ophthalmologist or another suitably qualified health care provider within the past 90 days prior to screening or in the period between screening and randomisation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (21):
- Japan (18):
  - Novo Nordisk Investigational Site, Adachi-ku, Tokyo
  - Novo Nordisk Investigational Site, Bunkyo-ku, Tokyo
  - Novo Nordisk Investigational Site, Chitose, Hokkaido
  - Novo Nordisk Investigational Site, Chuo-ku, Tokyo
  - Novo Nordisk Investigational Site, Chuo-ku,Tokyo
  - Novo Nordisk Investigational Site, Gunma
  - Novo Nordisk Investigational Site, Ibaraki
  - Novo Nordisk Investigational Site, Kanagawa
  - Novo Nordisk Investigational Site, Kashiwara-shi, Osaka
  - Novo Nordisk Investigational Site, Kobe, Hyogo
  - Novo Nordisk Investigational Site, Kumamoto
  - Novo Nordisk Investigational Site, Miyazaki
  - Novo Nordisk Investigational Site, Sapporo-shi, Hokkaido
  - Novo Nordisk Investigational Site, Shimotsuke-shi, Tochigi
  - Novo Nordisk Investigational Site, Suita-shi, Osaka
  - Novo Nordisk Investigational Site, Tokyo
  - Novo Nordisk Investigational Site, Toyama-shi, Toyama
  - Novo Nordisk Investigational Site, Yamato-shi, Kanagawa
- South Korea (3):
  - Novo Nordisk Investigational Site, Gyeonggi-do
  - Novo Nordisk Investigational Site, Seoul
  - Novo Nordisk Investigational Site, Yangsan

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://www.novonordisk-trials.com

REFERENCES:
- [Result] Davies M, Faerch L, Jeppesen OK, Pakseresht A, Pedersen SD, Perreault L, Rosenstock J, Shimomura I, Viljoen A, Wadden TA, Lingvay I; STEP 2 Study Group. Semaglutide 2.4 mg once a week in adults with overweight or obesity, and type 2 diabetes (STEP 2): a randomised, double-blind, double-dummy, placebo-controlled, phase 3 trial. Lancet. 2021 Mar 13;397(10278):971-984. doi: 10.1016/S0140-6736(21)00213-0. Epub 2021 Mar 2. PMID 33667417
- [Derived] Kadowaki T, Nishida T, Ogawa W, Overvad M, Tobe K, Yamauchi T. Effect of once-weekly subcutaneous semaglutide on abdominal visceral fat area in Japanese adults with overweight and obesity: A post hoc analysis of the STEP 6 trial. Obes Res Clin Pract. 2025 Mar-Apr;19(2):146-153. doi: 10.1016/j.orcp.2025.03.003. Epub 2025 Apr 4. PMID 40189961
- [Derived] Kadowaki T, Isendahl J, Khalid U, Lee SY, Nishida T, Ogawa W, Tobe K, Yamauchi T, Lim S; STEP 6 investigators. Semaglutide once a week in adults with overweight or obesity, with or without type 2 diabetes in an east Asian population (STEP 6): a randomised, double-blind, double-dummy, placebo-controlled, phase 3a trial. Lancet Diabetes Endocrinol. 2022 Mar;10(3):193-206. doi: 10.1016/S2213-8587(22)00008-0. Epub 2022 Feb 4. PMID 35131037

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 28 sites in 2 countries as follows (all sites screened and randomized):Japan (22 sites) and South korea (6 sites).
Pre-assignment Details: The trial has a 68-week treatment period (12 weeks of dose escalation and 56 weeks of maintenance dose for 1.7 milligram (mg) once weekly arm and 16 weeks of dose escalation and 52 weeks of maintenance dose for 2.4 mg once weekly arm). Participants were randomised in 4:1:2:1 ratio to receive either semaglutide subcutaneously (s.c.) 2.4 mg once-weekly, semaglutide placebo once-weekly, semaglutide s.c. 1.7 mg once-weekly or semaglutide placebo once-weekly.
Groups:
- Semaglutide 1.7 mg: Participants were to receive once-weekly s.c. injection of 0.25 mg semaglutide administered using a PDS290 pre-filled pen-injector with a 3 milliliter (mL) cartridge containing semaglutide 1.0 milligram per milliliter (mg/mL) or 3.0 mg/mL and followed a fixed-dose escalation regimen, with dose increases every 4 weeks (to doses of 0.5, 1.0 and 1.7 mg/week), aiming at reaching the maintenance dose of 1.7 mg once-weekly after 12 weeks. Treatment was continued on the maintenance dose of 1.7 mg once-weekly for an additional 56 weeks until week 68. The treatment was an adjunct to a reduced calorie diet and increased physical activity.
- Semaglutide 2.4 mg: Participants were to receive once-weekly s.c. injection of 0.25 mg semaglutide administered using a PDS290 pre-filled pen-injector with a 3 mL cartridge containing semaglutide 1.0 mg/mL or 3.0 mg/mL and followed a fixed-dose escalation regimen, with dose increases every 4 weeks (to doses of 0.5, 1.0, 1.7 and 2.4 mg/week), aiming at reaching the maintenance dose of 2.4 mg once-weekly after 16 weeks. Treatment was continued on the maintenance dose of 2.4 mg once-weekly for an additional 52 weeks until week 68. The treatment was an adjunct to a reduced calorie diet and increased physical activity.
- Placebo: Participants were to receive once-weekly s.c. injection of placebo matched to semaglutide for 68 weeks.
Period: Overall Study
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Started | 101 | 199 | 101
Full Analysis Set (FAS) | 101 | 199 | 101
Safety Analysis Set (SAS) | 100 | 199 | 101
Treated | 100 | 199 | 101
Completed | 99 | 195 | 101
Not Completed | 2 | 4 | 0
Not completed — Withdrawal by Subject | 2 | 4 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomised participants.
Groups:
- Semaglutide 1.7 mg: Participants were to receive once-weekly s.c. injection of 0.25 mg semaglutide administered using a PDS290 pre-filled pen-injector with a 3 mL cartridge containing semaglutide 1.0 mg/mL or 3.0 mg/mL and followed a fixed-dose escalation regimen, with dose increases every 4 weeks (to doses of 0.5, 1.0 and 1.7 mg/week), aiming at reaching the maintenance dose of 1.7 mg once-weekly after 12 weeks. Treatment was continued on the maintenance dose of 1.7 mg once-weekly for an additional 56 weeks until week 68. The treatment was an adjunct to a reduced calorie diet and increased physical activity.
- Total: Total of all reporting groups
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo | Total
Number analyzed (Participants) | 101 | 199 | 101 | 401
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51 (10) | 52 (12) | 50 (9) | 51 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 85 | 26 | 148
  Male | 64 | 114 | 75 | 253
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 101 | 199 | 101 | 401
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 101 | 199 | 101 | 401
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight (%)
Description: Change from baseline (week 0) in body weight for 'in-trial' observation period at week 68 is presented. In-trial observation period: the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0), week 68
Population: FAS which comprised all randomised participants. Overall Number of Participants Analyzed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage change
Groups:
- Semaglutide 1.7 mg: Participants were to receive once-weekly subcutaneous (s.c) injection of 0.25 mg semaglutide administered using a PDS290 pre-filled pen-injector with a 3 mL cartridge containing semaglutide 1.0 mg/mL or 3.0 mg/mL and followed a fixed-dose escalation regimen, with dose increases every 4 weeks (to doses of 0.5, 1.0 and 1.7 mg/week), aiming at reaching the maintenance dose of 1.7 mg once-weekly after 12 weeks. Treatment was continued on the maintenance dose of 1.7 mg once-weekly for an additional 56 weeks until week 68. The treatment was an adjunct to a reduced calorie diet and increased physical activity.
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 98 | 193 | 100
Percentage change | -9.9 (7.8) | -13.4 (8.6) | -1.9 (5.9)
Statistical Analysis 1: Comparison: Semaglutide 1.7 mg vs Placebo; Treatment policy estimand; Test type: Superiority; p < .0001, ANCOVA; Treatment difference = -7.52, 95% CI 2-sided [-9.62 to -5.43]
Statistical Analysis 2: Comparison: Semaglutide 2.4 mg vs Placebo; Treatment policy estimand; Test type: Superiority; p < .0001, ANCOVA; Treatment difference = -11.06, 95% CI 2-sided [-12.88 to -9.24]

2. Primary Outcome: Number of Participants Who Achieve (Yes/no): Body Weight Reduction More Than or Equal to 5%
Description: Number of participants who achieved greater than or equal to (≥) 5% weight loss at week 68 for in-trial observation period is presented. In the reported data, 'Yes' infers the number of participants who have achieved ≥ 5% weight loss, whereas 'No' infers the number of participants who have not achieved ≥ 5% weight loss. In-trial observation period: the uninterrupted time interval from the start of randomisation (week 0) to last trial-related subject-site contact (week 75).
Time Frame: At week 68
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 98 | 193 | 100
Participants
  Yes | 71 | 160 | 21
  No | 27 | 33 | 79
Statistical Analysis 1: Comparison: Semaglutide 1.7 mg vs Placebo; Treatment policy estimand; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 11.08, 95% CI 2-sided [5.53 to 22.22]
Statistical Analysis 2: Comparison: Semaglutide 2.4 mg vs Placebo; Treatment policy estimand; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 21.72, 95% CI 2-sided [11.27 to 41.86]

3. Secondary Outcome: Number of Participants Who Achieve (Yes/no): Body Weight Reduction More Than or Equal to 10%
Description: Number of participants who achieved greater than or equal to (≥) 10% weight loss at week 68 is presented. In the reported data, 'Yes' infers the number of participants who have achieved ≥ 10% weight loss, whereas 'No' infers the number of participants who have not achieved ≥ 10% weight loss. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomisation to last trial-related subject-site contact.
Time Frame: At week 68
Population: FAS which comprised all randomized participants. Overall number of participants analyzed = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 98 | 193 | 100
Participants
  Yes | 41 | 117 | 5
  No | 57 | 76 | 95

4. Secondary Outcome: Number of Participants Who Achieve (Yes/no): Body Weight Reduction More Than or Equal to 15%
Description: Number of participants who achieved greater than or equal to (≥) 15% weight loss at week 68 is presented. In the reported data, 'Yes' infers the number of participants who have achieved ≥ 15% weight loss, whereas 'No' infers the number of participants who have not achieved ≥ 15% weight loss. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomization to last trial-related subject-site contact.
Time Frame: At week 68
Population: FAS which comprised all randomised participants. Overall number of participants analyzed = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 98 | 193 | 100
Participants
  Yes | 24 | 79 | 3
  No | 74 | 114 | 97

5. Secondary Outcome: Number of Participants Who Achieve (Yes/no): Body Weight Reduction More Than or Equal to 20%
Description: Number of participants who achieved greater than or equal to (≥) 20% weight loss at week 68 is presented. In the reported data, 'Yes' infers the number of participants who have achieved ≥ 20% weight loss, whereas 'No' infers the number of participants who have not achieved ≥ 20% weight loss. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomisation to last trial-related subject-site contact.
Time Frame: At week 68
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 98 | 193 | 100
Participants
  Yes | 11 | 38 | 2
  No | 87 | 155 | 98

6. Secondary Outcome: Change in Waist Circumference Measured Midway Between the Lower Rib Margin and the Iliac Crest
Description: Change in waist circumference measured midway between the lower rib margin and the iliac crest from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomisation to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Centimeter (cm)
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 98 | 193 | 100
Centimeter (cm) | -7.8 (6.9) | -11.2 (7.5) | -1.8 (5.9)

7. Secondary Outcome: Change in Waist Circumference Measured According to the JASSO (Japan Society for the Study of Obesity) Guideline
Description: Change in Waist circumference measured according to the JASSO guideline from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomisation to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Centimeter (cm)
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 98 | 193 | 100
Centimeter (cm) | -7.6 (5.7) | -10.2 (6.8) | -1.9 (5.3)

8. Secondary Outcome: Change in Body Weight (Kg)
Description: Change in body weight from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomisation to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 98 | 193 | 100
Kilogram (kg) | -8.3 (6.1) | -11.3 (7.3) | -1.7 (5.6)

9. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Change in BMI from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomisation to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Kilogram per square meter (kg/m^2)
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 98 | 193 | 100
Kilogram per square meter (kg/m^2) | -3.1 (2.4) | -4.3 (2.8) | -0.6 (2.0)

10. Secondary Outcome: Change in Visceral Fat Area (VFA) (%)
Description: Change in VFA from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomisation to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: CT scan subpopulation included all randomised participants who had a CT scan assessment. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 45 | 86 | 43
Percentage change | -22.3 (31.3) | -41.0 (23.3) | -7.1 (19.5)

11. Secondary Outcome: Change in Visceral Fat Area (VFA) Centimeter Square (cm^2)
Description: as for outcome 10
Time Frame: Baseline (week 0) to week 68
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: centimeter square (cm^2)
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 45 | 86 | 43
centimeter square (cm^2) | -41.7 (47.0) | -67.4 (43.0) | -13.8 (38.6)

12. Secondary Outcome: Change in HbA1c (%)
Description: Change in glycosylated haemoglobin (HbA1c) from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomisation to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 98 | 193 | 100
Percentage of HbA1c | -0.9 (0.8) | -1.0 (1.0) | 0.0 (0.8)

13. Secondary Outcome: Change in HbA1c (mmol/Mol)
Description: as for outcome 12
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: millimoles per mole (mmol/mol)
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 98 | 193 | 100
millimoles per mole (mmol/mol) | -9.9 (8.9) | -10.6 (10.4) | -0.1 (8.3)

14. Secondary Outcome: Change in Fasting Plasma Glucose
Description: Change in fasting plasma glucose from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomization to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Milligrams per deciliter (mg/dL)
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 97 | 192 | 98
Milligrams per deciliter (mg/dL) | -18.3 (21.9) | -19.3 (22.6) | 1.7 (26.1)

15. Secondary Outcome: Change in Fasting Serum Insulin-ratio to Baseline
Description: Change in fasting serum insulin measured as milli-international units per milliliter (mIU/mL) from baseline (week 0) to week 68 is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomisation to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting serum insulin
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 97 | 190 | 98
Ratio of fasting serum insulin | 0.85 (65) | 0.71 (57.7) | 0.89 (49.4)

16. Secondary Outcome: Change in Systolic Blood Pressure
Description: Change in systolic blood pressure from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomisation to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 98 | 193 | 100
millimeters of mercury (mmHg) | -12 (13) | -11 (15) | -5 (15)

17. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Change in diastolic blood pressure from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomisation to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 98 | 193 | 100
mmHg | -5 (10) | -5 (10) | -3 (9)

18. Secondary Outcome: Change in Total Cholesterol-ratio to Baseline
Description: Change in total cholesterol measured as milligrams per deciliter (mg/dL) from baseline (week 0) to week 68 is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomisation to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 98 | 193 | 100
Ratio of total cholesterol | 0.93 (16.5) | 0.91 (13.3) | 1.00 (12.7)

19. Secondary Outcome: Change in High-density Lipoproteins (HDL)-Ratio to Baseline
Description: Change in HDL measured as milligrams per deciliter (mg/dL) from baseline (week 0) to week 68 is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomisation to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of high-density lipoproteins
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 98 | 193 | 100
Ratio of high-density lipoproteins | 1.06 (17.3) | 1.08 (13.7) | 1.06 (12.1)

20. Secondary Outcome: Change in Low-density Lipoproteins (LDL)-Ratio to Baseline
Description: Change in LDL measured as milligrams per deciliter (mg/dL) from baseline (week 0) to week 68 is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomization to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of low-density lipoproteins
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 98 | 193 | 99
Ratio of low-density lipoproteins | 0.90 (25.2) | 0.86 (23.5) | 0.95 (21.1)

21. Secondary Outcome: Change in Very Low-density Lipoproteins (VLDL)-Ratio to Baseline
Description: Change in VLDL measured as milligrams per deciliter (mg/dL) from baseline (week 0) to week 68 is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomization to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of very low-density lipoproteins
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 98 | 193 | 99
Ratio of very low-density lipoproteins | 0.79 (43.2) | 0.79 (43.2) | 1.05 (41.2)

22. Secondary Outcome: Change in Free Fatty Acids-ratio to Baseline
Description: Change in free fatty acids measured as milligrams per deciliter (mg/dL) from baseline (week 0) to week 68 is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomisation to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of free fatty acids
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 97 | 190 | 98
Ratio of free fatty acids | 1.04 (57.7) | 0.96 (59.1) | 1.28 (52.6)

23. Secondary Outcome: Change in Triglycerides-ratio to Baseline
Description: Change in triglycerides measured as milligrams per deciliter (mg/dL) from baseline (week 0) to week 68 is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomisation to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of triglycerides
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 98 | 193 | 99
Ratio of triglycerides | 0.78 (49.8) | 0.79 (43.8) | 1.05 (41.0)

24. Secondary Outcome: Change in High Sensitivity C-reactive Protein (hsCRP)-Ratio to Baseline
Description: Change in hsCRP measured in milligram per ilitre (mg/L) from baseline (week 0) to week 68 is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomisation to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of hsCRP
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 98 | 193 | 100
Ratio of hsCRP | 0.64 (218.3) | 0.39 (119.3) | 0.92 (123)

25. Secondary Outcome: Change in Plasminogen Activator Inhibitor-1 Activity-ratio to Baseline
Description: Change in plasminogen activator inhibitor-1 (PAI-1) activity measured in arbritary units per milliliter (AU/ml) from baseline (week 0) to week 68 is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomisation to last trial-related subject-site contact.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of PAI-1 activity
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 97 | 190 | 98
Ratio of PAI-1 activity | 0.83 (75.8) | 0.68 (62) | 1 (51.8)

26. Secondary Outcome: Change in Short Form 36 v2.0 Acute (SF-36) Score
Description: SF-36 is a 36-item patient-reported survey of patient health that measures participant's overall health-related quality of life (HRQoL). SF-36v2™ questionnaire measured eight domains of functional health and well-being as well as 2 component summary scores (physical component summary and mental component summary). This endpoint shows results for all the domains. The 0-100 scale scores from SF-36 were converted to norm-based scores to enable a direct interpretation in relation to distribution of scores in the 2009 U.S. general population. In metric of norm-based scores, 50 and 10 corresponds to mean and standard deviation respectively. Change from week 0 in domain scores and component summary scores were evaluated at week 68. A positive change score indicates an improvement since baseline. These endpoints were evaluated based on data from in-trial observation period which is uninterrupted time interval from randomisation to last contact with trial site.
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. Overall Number of Participants Analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 98 | 192 | 100
Score on a scale
  Change in SF-36:Physical functioning score | 0.0 (5.7) | 1.0 (3.7) | -0.5 (3.9)
  Change in SF-36: Role-Physical score | -1.6 (5.2) | -0.2 (4.7) | 0.3 (5.8)
  Change in SF-36: Bodily Pain score | -1.8 (9.2) | -1.1 (7.5) | -0.2 (8.8)
  Change in SF-36: General Health score | -1.4 (5.4) | 0.4 (5.8) | -0.6 (5.6)
  Change in SF-36: Vitality score | -2.4 (7.8) | -1.5 (6.8) | -0.9 (7.4)
  Change in SF-36: Social Functioning score | -0.8 (3.8) | -0.9 (6.2) | 0.3 (5.6)
  Change in SF-36: Role-Emotional score | -1.6 (5.6) | -1.1 (5.5) | -0.9 (4.1)
  Change in SF-36: Mental Health score | -1.9 (7.2) | -1.5 (6.7) | -1.2 (5.2)
  Change in SF-36: Physical component summary | -0.8 (6.0) | 0.7 (4.4) | 0.1 (5.3)
  Change in SF-36: Mental component summary | -2.0 (6.4) | -1.9 (6.4) | -1.0 (4.7)

27. Secondary Outcome: Change in Impact of Weight on Quality of Life-lite for Clinical Trials (IWQOL-Lite for CT) Score
Description: The Impact of Weight on Quality of Life Clinical Trials Version (IWQOL-Lite-CT) is designed to assess the impact of changes in weight on patients' quality of life within the context of clinical trials. IWQOL-Lite-CT is a 20-item questionnaire-based instrument used to assess the impact of body weight changes on participant's overall health-related quality of life (HRQoL). All IWQOL-Lite-CT composite scores range from 0 to 100, with higher scores reflecting better levels of functioning. This endpoint shows results for 'physical function score' physical and psychosocial domains, and for total'. The endpoint was evaluated based on the data from in-trial observation period which is the uninterrupted time interval from randomisation to last contact with trial site.
Time Frame: Baseline (week 0) to week 68
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 98 | 192 | 100
Score on a scale
  Physical function score | 2.6 (16.3) | 4.9 (15.1) | 0.5 (12.7)
  Physical | 1.9 (14.3) | 4.2 (14.4) | -0.8 (11.3)
  Psychosocial | 4.4 (11.9) | 5.2 (12.7) | -0.3 (12.1)
  Total | 3.5 (11.0) | 4.8 (11.8) | -0.5 (10.3)

28. Secondary Outcome: Number of Participants Who Achieve (Yes/no): Responder Definition Value for SF-36 Physical Functioning Score
Description: The number of participants experiencing a meaningful within participant improvement in SF-36 Physical function after 68 weeks was determined based on 3.7 threshold. The threshold of 3.7 is specific for overweight or obese population included in the study and calculated using patient global rating anchor questionnaires to reflect participants' own perspective based on Food and Drug Administration (FDA) recommendations. In the reported data, "Yes" infers the number of participants who have achieved an improvement in score greater than or equal to the threshold and "No" infers number of participants who have not achieved an improvement in score greater than or equal to the threshold. The endpoint was evaluated based on in-trial observation period which is the uninterrupted time interval from randomisation to last contact with trial site.
Time Frame: At week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 98 | 192 | 100
Participants
  Yes | 19 | 43 | 13
  No | 79 | 149 | 87

29. Secondary Outcome: Number of Participants Who Achieve (Yes/no): Responder Definition Value for IWQoL-Lite for CT Physical Function (5-items) Score
Description: The number of participants experiencing a meaningful within participant improvement in IWQOL-Lite-CT physical function after 68 weeks was determined based on thresholds of 14.6. The threshold of 14.6 is specific for the population with overweight or obesity included in the study and calculated using patient global rating anchor questionnaires to reflect participants' own perspective based on FDA recommendations. In the reported data, "Yes" infers the number of participants who have achieved an improvement in score greater than or equal to the threshold and "No" infers the number of participants who have not achieved an improvement in score greater than or equal to the threshold. The endpoint was evaluated based on in-trial observation period which is the uninterrupted time interval from randomisation to last contact with trial site.
Time Frame: At week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 98 | 192 | 100
Participants
  Yes | 19 | 49 | 11
  No | 79 | 143 | 89

30. Secondary Outcome: Number of Participants Who Achieved (Yes/no): HbA1c <7.0% (53 mmol/Mol)
Description: Number of participants who achieved HbA1c <7% (53 mmol/mol) at week 68 is presented. In the reported data, "Yes" infers the number of participants who have achieved HbA1c values less than the 7% and "No" infers the number of participants who have not achieved HbA1c values less than the 7%. The endpoint was evaluated based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomisation to last trial-related subject-site contact.
Time Frame: At week 68
Population: FAS included all randomised participants. Overall Number of Participants Analyzed = participants with type 2 diabetes at screening with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 25 | 49 | 25
Participants
  Yes | 24 | 43 | 1
  No | 1 | 6 | 24

31. Secondary Outcome: Number of Participants Who Achieved (Yes/no): HbA1c ≤6.5% (48 mmol/Mol)
Description: Number of participants who achieved HbA1c ≤6.5% (48 mmol/mol) at week 68 is presented. In the reported data, "Yes" infers the number of participants who have achieved HbA1c values less than or equal to 6.5% and "No" infers the number of participants who have not achieved HbA1c values less than or equal to 6.5%. The endpoint was evaluated based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomisation to last trial-related subject-site contact.
Time Frame: At week 68
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 25 | 49 | 25
Participants
  Yes | 22 | 40 | 1
  No | 3 | 9 | 24

32. Secondary Outcome: Number of Treatment-emergent AEs
Description: An adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a product, whether or not considered related to the product. All AEs mentioned here are treatment emergent adverse events (TEAE) defined as an event with onset during the on-treatment observation period. On-treatment observation period: the interval from the date of first trial product administration (week 0) to the date of last trial product administration (week 68) plus a 7 week follow-up period and excluding any off-treatment time intervals. Off-treatment time interval: time period with at least two consecutive missed doses.
Time Frame: Week 0 to week 75
Population: Safety analysis set (SAS) included all randomised participants exposed to at least one dose of randomised treatment.
Measure: Number; unit: Events
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 100 | 199 | 101
Events | 483 | 834 | 235

33. Secondary Outcome: Number of Serious Adverse Events
Description: A serious adverse event (SAE) is defined as any untoward medical occurrence that at any dose results in death, or is life-threatening, or requires inpatient hospitalization or causes prolongation of existing hospitalization results in persistent or significant disability/incapacity, or may have caused a congenital anomaly/birth defect, or requires intervention to prevent permanent impairment or damage. SAE results occurred from week 0 to week 75 is presented based on the on-treatment observation, which was defined as the interval from the date of first trial product administration (week 0) to the date of last trial product administration (week 68) plus a 7 week follow-up period and excluding any off-treatment time intervals. Off-treatment time interval: time period with at least two consecutive missed doses.
Time Frame: Week 0 to week 75
Population: Safety analysis set (SAS) included all randomised participants exposed to at least one dose of randomised treatment.
Measure: Number; unit: Events
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 100 | 199 | 101
Events | 10 | 12 | 7

34. Secondary Outcome: Number of Treatment Emergent Severe or Blood Glucose (BG) Confirmed Symptomatic Hypoglycaemia Episodes
Description: Hypoglycaemic episodes with onset during on-treatment observation period were considered treatment-emergent. Number of treatment emergent severe or BG confirmed symptomatic hypoglycaemia episodes with onset during on-treatment observation period were presented. Severe hypoglycaemia: episode requiring assistance of another person to administer carbohydrate, glucagon or take other corrective actions. plasma glucose (PG) concentrations may not be available during an event, but neurological recovery following return of PG to normal is considered sufficient evidence that event was induced by low PG concentration. BG confirmed symptomatic hypoglycaemia: episode that is BG confirmed by PG value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia. On-treatment observation period is interval from date of first trial product administration (week 0) to date of last trial product administration (week 68) plus 7-week follow-up period and excluding any off-treatment time intervals.
Time Frame: Week 0 to week 75
Population: Safety analysis set (SAS) included all randomised participants exposed to at least one dose of randomised treatment. Overall number of participants analyzed = participants with type 2 diabetes at screening.
Measure: Number; unit: Episodes
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 25 | 49 | 25
Episodes | 0 | 0 | 0

35. Secondary Outcome: Change in Pulse
Description: Change in pulse from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from on-treatment observation period, which was defined as the interval from the date of first trial product administration (week 0) to the date of last trial product administration (week 68) plus a 7 week follow-up period and excluding any off-treatment time intervals.
Time Frame: Baseline (week 0) to week 68
Population: SAS included all randomised participants exposed to at least one dose of randomised treatment. 'Overall Number of Participants Analysed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 93 | 186 | 98
Beats/minute | 6 (10) | 4 (9) | 2 (10)

36. Secondary Outcome: Change in Amylase: Ratio to Baseline
Description: Change in amylase measured in units/liter (U/L) from baseline (week 0) to week 68 is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment observation period, which was defined as the interval from the date of first trial product administration (week 0) to the date of last trial product administration (week 68) plus a 7 week follow-up period and excluding any off-treatment time intervals.
Time Frame: Baseline (week 0) to week 68
Population: as for outcome 35
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of amylase
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 93 | 186 | 98
Ratio of amylase | 1.09 (20.9) | 1.08 (23.2) | 0.93 (25.1)

37. Secondary Outcome: Change in Lipase: Ratio to Baseline
Description: Change in lipase measured in units/litre (U/L) from baseline (week 0) to week 68 is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment observation period, which was defined as the interval from the date of first trial product administration (week 0) to the date of last trial product administration (week 68) plus a 7 week follow-up period and excluding any off-treatment time intervals.
Time Frame: Baseline (week 0) to week 68
Population: as for outcome 35
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of lipase
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 93 | 186 | 98
Ratio of lipase | 1.56 (39.8) | 1.56 (45.4) | 0.96 (40.5)

38. Secondary Outcome: Change in Calcitonin: Ratio to Baseline
Description: Change in calcitonin measured in nanogram/litre (ng/L) from baseline (week 0) to week 68 is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment observation period, which was defined as the interval from the date of first trial product administration (week 0) to the date of last trial product administration (week 68) plus a 7 week follow-up period and excluding any off-treatment time intervals.
Time Frame: Baseline (week 0) to week 68
Population: as for outcome 35
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of calcitonin
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 93 | 186 | 98
Ratio of calcitonin | 0.98 (32.4) | 0.95 (34.6) | 0.94 (30.6)

39. Secondary Outcome: Change in QTCF Interval
Description: Change in QTCF Interval from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from on-treatment observation period, which was defined as the interval from the date of first trial product administration (week 0) to the date of last trial product administration (week 68) plus a 7 week follow-up period and excluding any off-treatment time intervals.
Time Frame: Baseline (week 0) to week 68
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: millisecond (msec)
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 92 | 186 | 96
millisecond (msec) | -2.2 (17.8) | -2.5 (15.2) | 5.6 (14.1)

ADVERSE EVENTS:
Time Frame: Week 0 to week 75.
Description: All presented AEs are treatment-emergent (i.e., TEAEs). Adverse events were defined as "treatment-emergent" (TEAE), if the onset of the event occurs in the on-treatment period. Results are based on the SAS which included all randomised participants exposed to at least one dose of randomised treatment.
Arm/Group | Semaglutide 1.7 mg | Semaglutide 2.4 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/199 | 0/101
Serious Adverse Events (participants affected / at risk) | 7/100 | 10/199 | 7/101
Other Adverse Events (participants affected / at risk) | 73/100 | 142/199 | 49/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 1.7 mg (N=100) | Semaglutide 2.4 mg (N=199) | Placebo (N=101)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bile duct adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis Meckel's (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rhegmatogenous retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 1.7 mg (N=100) | Semaglutide 2.4 mg (N=199) | Placebo (N=101)
Abdominal discomfort (Gastrointestinal disorders) | 11 (12) | 12 (16) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 7 (8) | 7 (8) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 12 (16) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (5) | 10 (13) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (10) | 5 (5) | 6 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (12) | 19 (20) | 9 (11)
Constipation (Gastrointestinal disorders) | 19 (22) | 52 (60) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 13 (13) | 0 (0)
Dental caries (Gastrointestinal disorders) | 4 (4) | 11 (12) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 22 (59) | 32 (52) | 6 (6)
Dizziness (Nervous system disorders) | 2 (4) | 14 (19) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 6 (17) | 9 (14) | 1 (4)
Gastroenteritis (Infections and infestations) | 7 (8) | 11 (13) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 10 (12) | 3 (3)
Nasopharyngitis (Infections and infestations) | 24 (36) | 53 (81) | 18 (24)
Nausea (Gastrointestinal disorders) | 18 (27) | 35 (66) | 4 (4)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 11 (13) | 9 (13)
Vomiting (Gastrointestinal disorders) | 10 (34) | 17 (29) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/74/NCT03811574/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/74/NCT03811574/SAP_001.pdf